CLINICAL TRIAL: NCT01572441
Title: Responses During Parent-child Interactions and Alcohol Use Behavior in Adolescents.
Brief Title: Parent-Adolescent Interactions and Adolescent Development
Acronym: PAIT
Status: Completed | Type: Observational
Sponsor: George Mason University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Tara M. Chaplin, Ph.D., Assistant Professor of Psychology, George Mason University
Other Study IDs: 0909005677; R01DA033431 (NIH)
Record Dates: First submitted 2012-04-03; First posted 2012-04-06 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Retain saliva sample.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 12-14 year olds: No intervention administered. This is a longitudinal observational study including observation of behaviors and physiological responses.

SUMMARY:
The purpose of this study is to observe parent-adolescent interactions and to examine the parenting behaviors and adolescent emotional and physiological responses that are associated with youth's substance use.

DETAILED DESCRIPTION:
The study examines parenting behaviors and adolescent emotional responses during parent-adolescent interactions and whether these predict youth's current and future substance use over a 3 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent between ages 12-14 years

Exclusion Criteria:

* For adolescent, Intelligence Quotient (IQ) < 70 on standardized test, for parent, evidence of inability to read or write.
* Evidence of a psychotic disorder for parent or adolescent
* Diagnosis of autism or pervasive developmental disorder for adolescent, as determined by parent report in the screening.
* For adolescent, current need for acute treatment of a psychiatric disorder, as determined by parent report in the study screening.
* For adolescent and parent, inadequate English proficiency to comprehend task instructions

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 12-14 year olds and their primary caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Substance Use | Baseline
  Measured by a combination of self-report on the Youth Risk Behavior Survey and the Teen Addiction Severity Index and urine toxicology and alcohol breathalyzer results.
Substance Use | 6 month follow-up
  Measured by a combination of self-report on the Youth Risk Behavior Survey and the Teen Addiction Severity Index and urine toxicology and alcohol breathalyzer results.
Substance Use | 1 year follow-up
  Measured by a combination of self-report on the Youth Risk Behavior Survey and the Teen Addiction Severity Index and urine toxicology and alcohol breathalyzer results.
Substance Use | 2 year follow-up
  Measured by a combination of self-report on the Youth Risk Behavior Survey and the Teen Addiction Severity Index and urine toxicology and alcohol breathalyzer results.
Substance Use | 3 year follow-up
  Measured by a combination of self-report on the Youth Risk Behavior Survey and the Teen Addiction Severity Index and urine toxicology and alcohol breathalyzer results.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Chaplin, Ph.D., Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale Stress Center, New Haven, Connecticut
  - George Mason University, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No
We will make data from the proposed laboratory study available to other researchers, after de-identifying study data and after publishing the main manuscripts on the study.

REFERENCES:
- [Background] Chaplin TM, Sinha R, Simmons JA, Healy SM, Mayes LC, Hommer RE, Crowley MJ. Parent-adolescent conflict interactions and adolescent alcohol use. Addict Behav. 2012 May;37(5):605-12. doi: 10.1016/j.addbeh.2012.01.004. Epub 2012 Jan 13. PMID 22341765
- [Result] Turpyn CC, Chaplin TM, Cook EC, Martelli AM. A person-centered approach to adolescent emotion regulation: Associations with psychopathology and parenting. J Exp Child Psychol. 2015 Aug;136:1-16. doi: 10.1016/j.jecp.2015.02.009. Epub 2015 Apr 4. PMID 25846016